CLINICAL TRIAL: NCT00748085
Title: A Multi-Center Study of CryoSpray Ablation(tm)in Malignant Airway Disease to Determine, Safety, and Tissue Effect in the Lung (ICE the MAD)
Brief Title: CryoSpray Ablation(tm)in Malignant Airway Disease to Determine Safety, and Tissue Effect in the Lung (ICE the MAD)
Acronym: ICEtheMAD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Business Reasons
Sponsor: CSA Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-0106
Record Dates: First submitted 2008-09-04; First posted 2008-09-08 (Estimated); Results first posted 2014-07-16 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-06

CONDITIONS: Lung Cancer; Mesothelioma
Keywords: Malignant Airway Disease; Lung Cancer; Inoperable Lung Cancer; Mesothelioma; Endoluminal Tumor
MeSH Terms: conditions — Lung Neoplasms; Mesothelioma | interventions — Drug Delivery Systems; Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cryospray Ablation (Experimental): Cryospray Ablation 4, 5-second spray cycles
  Interventions: Device: CryoSpray Ablation

INTERVENTIONS:
Device: CryoSpray Ablation — Treatment dosimetry will be up to 4, 5-second spray cycles. Subjects will have initial cryospray treatment. Subjects may undergo up to one bronchoscopy with CryoSpray Ablation every seven days for a total of four (4) treatments in the first month.
  Other Names: CryoSpray Ablation(TM)System; CSA (TM) System; Cryo Spray Therapy; CSA; Cryotherapy; Cryo Spray Ablation

SUMMARY:
The purpose of this study is to evaluate the safety, and tissue effect of the CryoSpray Ablation(TM) System (CryoSpray Ablation(TM), "CSA" or "cryospray therapy") at multiple centers to treat malignant airway disease in the lung using liquid nitrogen sprayed through a catheter via flexible fiber optic bronchoscopy (FFB)

DETAILED DESCRIPTION:
The primary endpoint is efficacy of the cryogen on the tumor evaluated by histopathological data and visual inspection along with visual confirmation of an absence of scarring and stricturing of the airway. The primary safety endpoint is the reporting of all adverse events. The primary symptom measures are the St. Georges Respiratory Questionnaire (SGRQ) and the Borg Dyspnea Index (BDI).

The secondary endpoint will consist of a measure of treatment efficacy and improvement in luminal patency assessed by visual inspection. If after the initial repeat bronchoscopy, the investigator determines that there is no immediate need for further intervention, then any future bronchoscopy will be performed upon the subject presenting with symptoms.

The proposed study will take place at up to three centers consisting of up to a total of 30 subjects with malignant airway obstruction. Treatment dosimetry will be up to 4, 5-second spray cycles. Subjects will have initial cryospray treatment at Day 0. Subjects will undergo repeat bronchoscopy in the first seven days after the initial treatment to check for mucosal sloughing and to reassess luminal patency of the airway. Subjects may undergo up to one bronchoscopy with CSA therapy every seven days for a total of four (4) treatments in the first month. If they present with symptoms thereafter, then a repeat bronchoscopy will be performed; if luminal obstruction is noted, then the subject will begin the treatment protocol again. Subjects may also have rigid/flexible bronchoscopy with laser or electrocautery snare for debulking of tumors. If disease exists bilaterally, only one side will be sprayed initially.

The study population consists of up to 30 subjects with malignant airway obstruction as a consequence of an endoluminal tumor that obstructs a portion of the respiratory tree below the vocal chords. These subjects will have been apprised of Standard of Care options, and will have rejected those options or have been deemed ineligible for them. Subjects must have a signed consent form and satisfy all study inclusion and exclusion criteria.

It is estimated that enrollment will take approximately 6 months. Each subject will receive CryoSpray treatments over the course of 1 year.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or greater
* Deemed a candidate for cryotherapy based on physician physical or medical history review
* Deemed inoperable based on institutional criteria.

Exclusion Criteria:

* Pregnant or nursing
* Planning to sire a child while enrolled in the study
* Known history of unresolved drug or alcohol dependency that would limit ability to comprehend or follow instructions related to informed consent, post-treatment instructions, or follow-up guidelines.
* Refusal or inability to give consent.
* Concurrent induction chemotherapy.
* Radiation therapy within the last 30 days which involved the any area between the vocal chords and the diaphragm.
* Medical contraindication or potential problem that would preclude study participation
* Concurrent participation in other experimental studies
* Uncontrolled coagulopathy or bleeding diathesis
* Serious medical illness, including:
* Uncontrolled congestive heart failure;
* Uncontrolled angina;
* Myocardial infarction;
* Cerebrovascular accident within 6 months prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-10; Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William S Krimsky, M.D., Principal Investigator — Franklin Square Hospital Center
Locations (1):
- Franklin Square Hospital Center, Baltimore, Maryland, United States

REFERENCES:
- [Background] Johnston CM, Schoenfeld LP, Mysore JV, Dubois A. Endoscopic spray cryotherapy: a new technique for mucosal ablation in the esophagus. Gastrointest Endosc. 1999 Jul;50(1):86-92. doi: 10.1016/s0016-5107(99)70352-4. PMID 10385730
- [Background] Ell C, May A, Gossner L, Pech O, Gunter E, Mayer G, Henrich R, Vieth M, Muller H, Seitz G, Stolte M. Endoscopic mucosal resection of early cancer and high-grade dysplasia in Barrett's esophagus. Gastroenterology. 2000 Apr;118(4):670-7. doi: 10.1016/s0016-5085(00)70136-3. PMID 10734018
- [Background] Champion G, Richter JE, Vaezi MF, Singh S, Alexander R. Duodenogastroesophageal reflux: relationship to pH and importance in Barrett's esophagus. Gastroenterology. 1994 Sep;107(3):747-54. doi: 10.1016/0016-5085(94)90123-6. PMID 8076761
- [Background] Eisen GM, Sandler RS, Murray S, Gottfried M. The relationship between gastroesophageal reflux disease and its complications with Barrett's esophagus. Am J Gastroenterol. 1997 Jan;92(1):27-31. PMID 8995932
- [Background] Johnston MH. Cryotherapy and other newer techniques. Gastrointest Endosc Clin N Am. 2003 Jul;13(3):491-504. doi: 10.1016/s1052-5157(03)00044-8. PMID 14629105
- [Background] Cash BD, Johnston LR, Johnston MH. Cryospray ablation (CSA) in the palliative treatment of squamous cell carcinoma of the esophagus. World J Surg Oncol. 2007 Mar 16;5:34. doi: 10.1186/1477-7819-5-34. PMID 17367523
- [Background] Field JK, Youngson JH. The Liverpool Lung Project: a molecular epidemiological study of early lung cancer detection. Eur Respir J. 2002 Aug;20(2):464-79. doi: 10.1183/09031936.02.00290202. PMID 12212983
- [Background] Pinsonneault C, Fortier J, Donati F. Tracheal resection and reconstruction. Can J Anaesth. 1999 May;46(5 Pt 1):439-55. doi: 10.1007/BF03012943. PMID 10349923
- [Background] Dumot JA. Cryotherapy Ablation for Esophageal HGD or IMCA in High Risk, Non-Surgical Patients. DDW2007 Abstract submission. Cleveland Clinic Foundation (pending publication)
- [Background] Greenwald BD. CryoSpray Ablation of Early Esophageal Cancer. DDW 2007 Abstract submission. University of Maryland Medical Center. (pending publication)
- [Background] Johnston M, Horwhat J, Dubois A, Schoenfeld P. Endoscopic cryotherapy in the swine esophagus: A follow-up study (Abstract). Gastrointestinal Endoscopy 49:AB126, 1999.
- [Background] Johnston MH, Horwhat JD, Haluska, Moses FM. Depth of injury following endoscopic spray cryotherapy: EUS assisted evaluation of mucosal ablation and subsequent healing in the swine model (Abstract). Gastrointestinal Endoscopy 51: AB98, 3462, 2000.
- [Background] Johnston MH. Endoscopic cryotherapy: A new ice age in gastroenterology? Medscape Gastroenterology 2: 187, 2000.
- [Background] Eastone JA, Horwhat D, Haluska O, Mathews J, Johnston M. Cryoablation of swine esophageal mucosa: A direct comparison to argon plasma coagulation (APC) and multipolar electrocoagulation (MPEC) [Abstract] Gastrointestinal Endoscopy 53: A3448, 2001.
- [Background] Johnston MH, Eastone JA, Horwhat JD. Reversal of Barrett's esophagus with cryotherapy [Abstract]. American Journal of Gastroenterology 98(9 Suppl): A30, S11, 2003.
- [Background] Johnston MH, Cash BD, Horwhat JD, Johnston LR, Dykes CA, Mays HS. Cryoablation of Barrett's Esophagus (BE) [Abstract]. Gastroenterology 130 (4, Suppl.2): A640, 2006.
- [Background] Johnston MH, Cash BD, Dykes CA, Mays HS, Johnston LR. Cryoablation of dysplasia in Barrett's Esophagus (BE) and early stage esophageal cancer [Abstract]. Gastrointestinal Endoscopy 63 (5): April, 2006.
- [Background] Johnston MH, Eastone JA, Horwhat JD, Cartledge J, Mathews JS, Foggy JR. Cryoablation of Barrett's esophagus: a pilot study. Gastrointest Endosc. 2005 Dec;62(6):842-8. doi: 10.1016/j.gie.2005.05.008. PMID 16301023

RESULTS

PARTICIPANT FLOW:
Groups:
- 1-all Subjects: CryoSpray Ablation (TM) System: Treatment dosimetry will be up to 4, 5-second spray cycles. Subjects will have initial cryospray treatment at Day 0. Subjects will undergo repeat bronchoscopy in the first seven days after the initial treatment to check for mucosal sloughing and to reassess luminal patency of the airway. Subjects may undergo up to one bronchoscopy with CSA therapy every seven days for a total of four (4) treatments in the first month. If they present with symptoms thereafter, then a repeat bronchoscopy will be performed; if luminal obstruction is noted, then the subject will begin the treatment protocol again. Subjects may also have rigid/flexible bronchoscopy with laser or electrocautery snare for debulking of tumors. If disease exists bilaterally, only one side will be sprayed initially.
Period: Overall Study
Arm/Group | 1-all Subjects
Started | 5
Completed | 5 (No analysis -study terminated for business reasons.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 1-all Subjects
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of the Cryogen on a Tumor Evaluated by Histopathological Data and Visual Inspection Along With Visual Confirmation of Absence of Scarring and Stricturing of the Airway. The Primary Safety Endpoint is the Reporting of All Adverse Events.
Time Frame: 1 year
Population: no analysis conducted-study terminated for business reasons
Arm/Group | 1-all Subjects
Number analyzed (Participants) | 0

2. Secondary Outcome: Consists of a Measure of Treatment Efficacy and Improvement in Luminal Patency Assessed by Visual Inspection.
Time Frame: 1 year
Population: no analysis conducted. Study terminated for business reasons
Arm/Group | 1-all Subjects
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | 1-all Subjects
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 1/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1-all Subjects (N=5)
Vertigo (Ear and labyrinth disorders) | 1 (1)
chest pain (Cardiac disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
other-Hoarseness (Ear and labyrinth disorders) | 1 (1)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No